CLINICAL TRIAL: NCT05211375
Title: Comparisons of Metabolic Effect of Sleeve Gastrectomy With Duodenojejunal Bypass and Sleeve Gastrectomy (MEDUSA): A Multicenter Randomized Controlled Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ajou University School of Medicine (Other); The Catholic University of Korea (Other); The Catholic University of Korea Eunpyeong St. Mary's Hospital (Unknown); Ewha University Seoul Hospital (Unknown); Seoul Metropolitan Boramae Hospital (Unknown); Soonchunhyang University Hospital (Other); Korea University (Other)
Responsible Party: Principal Investigator, Young Suk Park, MD, Principle Investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDUSA
Record Dates: First submitted 2022-01-04; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2; Bariatric Surgery; Surgical Procedures, Operative; Asians
Keywords: Bariatric Surgery; Metabolic Surgery; Diabetes Remission
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SG group (Active Comparator): Patients undergoing sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- DJB group (Experimental): Patients undergoing duodenojejunal bypass with sleeve gastrectomy
  Interventions: Procedure: Duodenojejunal bypass

INTERVENTIONS:
Procedure: Duodenojejunal bypass — Sleeve gastrectomy will be performed in the same manner as in the SG group. DJB will be performed by transection of the duodenum and bypassing 250 cm of the proximal jejunum. The handsewn suture will be used for duodenojejunal anastomosis, and the size of anastomosis will be 1.5 - 2 cm. Single anastomosis will be performed rather than Roux-en-Y fashion.
  Arms: DJB group
Procedure: Sleeve gastrectomy — Sleeve gastrectomy will be performed using 36-38 Fr bougie. The initial stapling start point will be between 4-6 cm from the pylorus, and the last stapling will be performed at least 1 cm away from His angle. The height of the automatic stapler will be selected based on the researcher's discretion.
  Arms: SG group

SUMMARY:
In this study, the effects of SG with DJB and SG alone for the treatment of type 2 diabetes mellitus (T2DM) will be compared in patients other than the two groups at both extremes who are expected to show excellent effects of metabolic surgery with SG alone (mild T2DM) and who need SG with DJB (severe T2DM).

This study is to target patients with poor blood sugar control despite current medical treatment, although the beta-cell function of the pancreas is preserved. Therefore, this study is aimed at patients who have been using insulin for less than 10 years with T2DM, or taking diabetic medications with HbA1c ≥ 7.0% for less than 10 years with T2DM.

The investigators hypothesize that the treatment effects of SG with DJB for T2DM will be superior to that of SG in this group

DETAILED DESCRIPTION:
Most Asian patients undergoing metabolic surgery for the treatment of T2DM have BMI as low as 30-35 kg/m2. If SG is performed for the treatment of T2DM in these patients, weight may decrease after the surgery; however, T2DM may recur after 6 months to 1 year. Therefore, it is difficult to find clinical studies on SG for metabolic surgery in Asians, and gastric bypass may be more appropriate as metabolic surgery. However, gastroscopy for the remnant stomach after gastric bypass is practically impossible. Therefore, gastric bypass may be a fatal drawback for East Asian patients with a high incidence of gastric cancer. In recent years, modified duodenal switch (SG with duodenojejunal bypass [DJB], which is defined as the procedure that makes jejunal bypass shorter than the traditional duodenal switch) is often performed as metabolic surgery, and studies on this surgical technique are being actively conducted in Japan.

SG with DJB has both effects of stomach restriction and foregut bypass. However, SG with DJB is more disadvantageous compared to SG alone in nutrient absorption after surgery. This is a natural result of bypassing the duodenum and proximal jejunum. Therefore, SG with DJB should not be performed when it is unnecessary, and it should be performed in patients who are expected to show significant improvement in T2DM. However, there is no existing guideline on which patients can receive SG with DJB or SG alone, and there are also no clinical studies on these aspects.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* BMI equal to or greater than 27.5 kg/m2
* T2DM duration ≤ 10 years
* Using insulin, or HbA1c ≥ 7.0% while taking diabetes medication
* C-peptide level higher than 1.0 ng/mL
* Presence of type 2 diabetes fulfilling the following criteria
* Consent to not become pregnant for at least 1 year after surgery
* Willingness to provide voluntary informed consent

Exclusion Criteria:

* Presence of uncontrolled severe gastroesophageal reflux (LA classification C or more in esophagogastroduodenoscopy)
* History of previous metabolic surgery for T2DM
* History of gastrointestinal surgery, such as gastrectomy or anti-reflux surgery, which may affect the result of metabolic surgery
* Therapy regimen of more than 3 psychiatric drugs owing to poorly controlled psychiatric disorders
* Suicidal attempts within the last 12 months
* Treatment for alcohol and drug abuse within the last 12 months
* Vulnerability factors (lacking mental capacity, pregnancy or planning of pregnancy, lactation)
* Unsuitability as per the discretion of the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2031-01-03 (Estimated); Study Completion 2036-01-03 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate of type 2 diabetes | 5 years after surgery
  HbA1c <6% (or fasting blood glucose [FBG] <100 mg/dL) without using any diabetes medication

SECONDARY OUTCOMES:
Complete remission rate of type 2 diabetes | 1, 3, 10 years after surgery
  HbA1c <6% (or fasting blood glucose [FBG] <100 mg/dL) without using any diabetes medication
Partial remission rate of type 2 diabetes | 1, 3, 5, 10 years after surgery
  Definition of partial remission of diabetes: HbA1c of 6-6.4% (or FBG of 100-125 mg/dL) without using any diabetes medication
Improvement rate of type 2 diabetes | 1, 3, 5, 10 years after surgery
  Definition of improvement of diabetes: Significant reduction in HbA1c (or FBG) level or decrease in the number of diabetic drugs or stoppage of insulin that does not meet the definition of remission.
Hypertension remission rate | 1, 3, 5, 10 years after surgery
  Definition of complete remission of hypertension: Blood pressure (BP) <120/80 mmHg without taking BP medication Definition of partial remission of hypertension: BP of 120-140/80-89 mmHg without taking BP medication
Hypertension improvement rate | 1, 3, 5, 10 years after surgery
  Definition of improvement of hypertension: Decrease in the number or dose of BP medications or decreased BP while taking medication
Hyperlipidemia remission rate | 1, 3, 5, 10 years after surgery
  Definition of remission of hyperlipidemia: Normal lipid profile (triglyceride [TG] <150 mg/dL and low-density lipoprotein [LDL] of 129 mg/dL or less and high-density lipoprotein [HDL] of 40 mg/dL or above) without taking hyperlipidemic drugs
Hyperlipidemia improvement rate | 1, 3, 5, 10 years after surgery
  Definition of improvement of hyperlipidemia: Reduced number or dose of hyperlipidemic drugs or improved lipid profile while taking hyperlipidemic drugs
Prevalence of GERD | 1, 3, 5, 10 years after surgery
  Acid reflux symptoms and positive endoscopic findings (LA classification A or more)
Trace element deficiency rate (iron, vitamin B12, folate, vitamin B1, vitamin D, copper [Cu], and zinc [Zn]) | 1, 3, 5, 10 years after surgery
  Iron deficiency: ferritin <20 ng/mL or iron <50 mcg/dL Vitamin B12 deficiency: <200 pg/mL, vitamin B12 suboptimal: 200 - <400 pg/mL Folate deficiency: <10nmol/L (4.4ng/mL) Vitamin B1 deficiency: <2.36 mcg/dL Vitamin D deficiency: <20 mg/mL, vitamin D insufficiency: 20-<30 ng/mL Cu deficiency: <75 mcg/dL Zn deficiency: <70 mcg/dL in women, < 74 mcg/dL in men
Changes in body weight | 1, 3, 5, 10 years after surgery
  kilograms
Changes in body composition | 1, 3, 5, 10 years after surgery
  body fat percentage(%), body fat mass (kg), and muscle mass(kg)
Changes in Quality of life | 1, 3, 5, 10 years after surgery
  IWQOL-Lite, SF-12
Early complication rate | Early: within 30 days after surgery
Late complication rate | Late: later than 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Young Suk Park, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofso D, Fatima F, Borgeraas H, Birkeland KI, Gulseth HL, Hertel JK, Johnson LK, Lindberg M, Nordstrand N, Cvancarova Smastuen M, Stefanovski D, Svanevik M, Gretland Valderhaug T, Sandbu R, Hjelmesaeth J. Gastric bypass versus sleeve gastrectomy in patients with type 2 diabetes (Oseberg): a single-centre, triple-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2019 Dec;7(12):912-924. doi: 10.1016/S2213-8587(19)30344-4. Epub 2019 Oct 31. PMID 31678062
- [Background] Aminian A, Brethauer SA, Andalib A, Nowacki AS, Jimenez A, Corcelles R, Hanipah ZN, Punchai S, Bhatt DL, Kashyap SR, Burguera B, Lacy AM, Vidal J, Schauer PR. Individualized Metabolic Surgery Score: Procedure Selection Based on Diabetes Severity. Ann Surg. 2017 Oct;266(4):650-657. doi: 10.1097/SLA.0000000000002407. PMID 28742680
- [Background] Brethauer SA, Kim J, el Chaar M, Papasavas P, Eisenberg D, Rogers A, Ballem N, Kligman M, Kothari S; ASMBS Clinical Issues Committee. Standardized outcomes reporting in metabolic and bariatric surgery. Surg Obes Relat Dis. 2015 May-Jun;11(3):489-506. doi: 10.1016/j.soard.2015.02.003. No abstract available. PMID 26093765